CLINICAL TRIAL: NCT06177327
Title: Screening and Epidemiology of Hepato-pancreato-biliary Abnormalities in Fibrous Dysplasia of Bone /McCune Albright Syndrome: the TIM-DYS Study
Brief Title: Hepato-pancreato-biliary Abnormalities in Fibrous Dysplasia of Bone/McCune Albright Syndrome
Acronym: TIM-DYS
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 23-5288
Record Dates: First submitted 2023-12-11; First posted 2023-12-20 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Fibrous Dysplasia of Bone
Keywords: Fibrous dysplasia of bone; McCune Albright syndrome; pancreatic neoplasms; IPMN
MeSH Terms: conditions — Fibrous Dysplasia of Bone; Fibrous Dysplasia, Polyostotic; Pancreatic Neoplasms | interventions — Mass Screening

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults with polyostotic fibrous dysplasia McCune Albright syndrome: A retrospective data collection and statistical analyses will be performed. Adults with polyostotic fibrous dysplasia McCune Albright syndrome, who underwent an hepato-bilio-pancreatic MRI since January 2002, during their follow-up
  Interventions: Other: Screening for hepato-bilio-pancreatic abnormalities in Fibrous dysplasia of bone /McCune Albright syndrome , description and characterization of the lesions.

INTERVENTIONS:
Other: Screening for hepato-bilio-pancreatic abnormalities in Fibrous dysplasia of bone /McCune Albright syndrome , description and characterization of the lesions. — Data collection from hepato-bilio-pancreatic Magnetic Resonance Imaging realized during the follow up of patients with Fibrous dysplasia of bone /McCune Albright syndrome

SUMMARY:
Fibrous dysplasia of bone /McCune Albright syndrome (FD/MAS) is a rare bone disease caused by somatic mutations in GNAS gene. This GNAS mutation predisposes to cancers, including breast cancer, thyroid cancer, chondrosarcoma and osteosarcoma, as well as biliary tract anomalies, liver-tumors or pancreatic tumors - IPMNs. Intraductal papillary and mucinous neoplasms of the pancreas (IPMN) are cystic intraepithelial ductal lesions developed at the expense of pancreatic ducts. They are pre-cancerous lesions, requiring monitoring and, in case of progression or malignant degeneration, surgical resection. Pancreatic MRI screening of patients with polyostotic FD and MAS is recommended.

The aim of this study is to investigate the epidemiology and characteristics of these hepato-pancreato-biliary abnormalities (prevalence, age of onset, degeneration), based on magnetic resonance imaging (MRI) realized during the follow-up of patients with FD/MAS treated in a French FD expert center.

A better understanding of these IPMNs and other digestive abnormalities will enable clinicians to improve the management and monitoring in this high-risk population.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years with polyostotic FD/MAS
* Followed up in the national FD reference center (Lyon) or in a FD French expert center: Angers, Bordeaux, Brest, Caen, Clermont-Ferrand, Lille, Marseille, Montpellier, Nice, Paris, Poitiers, Rennes, Saint-Etienne, Strasbourg.
* who had an hepato-bilio-pancreatic MRI during their follow-up, since January 2002
* No objection to data collection

Exclusion Criteria:

-Opposition to data collection

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 545 (Estimated)
Dates: Start 2024-01-19 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-12-12 (Estimated)

PRIMARY OUTCOMES:
Describe hepato-bilio-pancreatic abnormalities in FD/MAS and estimate the prevalence of IPMN. | hepato-bilio-pancreatic MRI performed from January 2002 until December 2024.
  Hepato-bilio-pancreatic abnormalities (size, number, complications) will be described based on hepato-bilio-pancreatic MRI.

CONTACTS AND LOCATIONS:
Locations (16):
- France (16):
  - CHU Angers, Angers
  - Groupe Hospitalier Pellegrin - Chu, Bordeaux
  - CHU de Brest - Hôpital de la Cavale Blanche, Brest
  - Chu de Caen Normandie, Caen
  - Chu de Clermont-Ferrand, Clermont-Ferrand
  - Chu de Lille, Lille
  - Service Rhumatologie, pavillon F Hopital E. Herriot, Lyon
  - Assistance Publique - Hopitaux de Marseille (Ap-Hm, Marseille
  - Chu de Montpellier, Montpellier
  - CHU de Nice, Nice
  - Assistance Publique - Hopitaux de Paris (Ap-Hp), Paris
  - CHU de Poitiers, Poitiers
  - Chu de Rennes, Rennes
  - Chu de Saint-Etienne, Saint-Etienne
  - Hopitaux Universitaires de Strasbourg, Strasbourg
  - Chu de Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No